CLINICAL TRIAL: NCT01326481
Title: An Open Label Phase 1B Dose-Finding Study of TRC105 in Combination With Capecitabine for Progressive or Recurrent Metastatic Breast Cancer
Brief Title: Open Label Dose-Finding Study of TRC105 Plus Capecitabine for Metastatic Breast Cancer
Acronym: TRC105
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Collaborators: Roswell Park Cancer Institute (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105BC102
Record Dates: First submitted 2011-03-25; First posted 2011-03-31 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Breast Cancer
Keywords: TRC105; Breast Cancer; CD105; Endoglin; TRACON Pharma; Roswell Park Cancer Institute; Department of Defense
MeSH Terms: conditions — Breast Neoplasms | interventions — carotuximab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single (Experimental): All patients received TRC105 + capecitabine
  Interventions: Drug: TRC105; Drug: Capecitabine

INTERVENTIONS:
Drug: TRC105 — IV
  Other Names: carotuximab
Drug: Capecitabine — oral
  Other Names: xeloda

SUMMARY:
The purpose of this study is to determine the recommended phase 2 dose and overall safety and tolerability of TRC105 when given in combination with capecitabine for the treatment of patients with progressive or recurrent metastatic breast cancer.

DETAILED DESCRIPTION:
All patients were required to sign a consent form prior to undertaking any study-related procedures. Prospective patients were screened to determine if they qualified for the study within 28 days of enrollment. Patients who qualified received TRC105 i.v. over 1 to 4 hours on Day 1, Day 4, Day 8 and Day 15 of the initial 21-day cycle and Day 1, Day 8 and Day 15 of every subsequent 21-day cycle in combination with 1000 mg/m2 capecitabine BID for 14 days of each 21-day cycle. Those who tolerated TRC105 without any infusion reactions were eligible for reduced infusion durations. After 3 cycles of treatment, patients who demonstrated a response of complete response (CR), partial response (PR) or stable disease (SD) were eligible for additional treatment for up to six months (9 total cycles). Upon discussion with TRACON, patients judged by the Principal Investigator to be benefiting from treatment were able to continue treatment on this protocol beyond six months.

Toxicities were graded according to the NCI CTCAE Version 4.0. Patients who exited the study for reasons other than drug-related toxicity prior to completion of the first 21-day cycle were replaced. Intra-patient dose escalation was not allowed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven advanced solid cancer for which curative therapy is not available (Part 1 only)
* Histologically proven metastatic Her-2-negative breast cancer (Part 2 only)
* Measurable disease by RECIST 1.1 criteria (Part 2 only)
* Willing and able to consent for self to participate in study
* Progressive or recurrent disease after prior systemic chemotherapy regimen
* Age ≥ 18 years
* ECOG performance status of 0 or 1
* Resolution of all acute toxic effects of prior therapy to NCI CTCAE Grade ≤ 1 or baseline (except alopecia)
* Adequate organ function

Exclusion Criteria:

* Prior treatment with more than one systemic chemotherapy regimen for metastatic disease.
* Prior treatment with TRC105
* History of hypersensitivity reaction to antimetabolite therapy
* Receipt of an investigational agent within 28 days of starting study treatment
* Prior surgery (including open biopsy), radiation therapy or systemic therapy within 28 days of starting study treatment
* Minor surgical procedures within 14 days prior to first dose of TRC105
* History of brain metastasis, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease
* Angina, MI, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, pulmonary embolism, DVT, PTCA or CABG within the past 6 months
* Uncontrolled chronic hypertension defined as systolic > 140 or diastolic > 90 despite optimal therapy
* Past medical history of acquired or inherited coagulopathy including patients with known hereditary hemorrhagic telangiectasia
* Thrombolytic or anticoagulant use (except to maintain i.v. catheters) within 10 days prior to first dose with TRC105
* Cardiac dysrhythmias of NCI CTCAE Grade ≥ 2 within the last month
* Hemorrhage within 28 days of starting study treatment
* Unhealed wounds within 28 days of starting study treatment
* History of peptic ulcer disease or gastritis within the past 6 months, unless treated for the condition and complete resolution has been documented by esophagogastroduodenoscopy (EGD) within 28 days of starting study treatment
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
* Known active viral or nonviral hepatitis
* History of hypersensitivity reaction to human or mouse antibody products
* Lung cancer with central chest lesions
* Pregnancy or breastfeeding

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-06; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Theuer, MD PhD, Study Chair — Tracon Pharmaceuticals Inc.
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Roswell Park Cancer Institute, Buffalo, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Carotuximab (TRC105) Plus Capecitabine: All patients received TRC105 + capecitabine
  TRC105: IV (7.5 or 10 mg/kg weekly)
  Capecitabine: oral (1,000 mg/m2 BID)
Period: 7.5 mg/kg TRC105, 1000 mg/m2 Cape
Arm/Group | Carotuximab (TRC105) Plus Capecitabine
Started | 4
Completed | 3
Not Completed | 1
Not completed — Adverse Event | 1
Period: 10 mg/kg TRC105, 1000 mg/m2 Cape
Arm/Group | Carotuximab (TRC105) Plus Capecitabine
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients who received at least a portion of a dose of TRC105
Groups:
- Single: All patients received TRC105 + capecitabine TRC105: IV (7.5 or 10 mg/kg weekly) Capecitabine: oral (1,000 mg/m2 BID)
Arm/Group | Single
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants] — Age at the time of enrollment
  Participants
    <=18 years | 0
    Between 18 and 65 years | 15
    >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 53 [33 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Determine Maximum Tolerated Dose of TRC105 in Combination With Capecitabine
Description: Assess safety and dose limiting toxicity by dose cohort and coding all terms utilized MedDRA version 14.1.
Time Frame: 1.5 years
Population: All patients who received at least a portion of a dose of TRC105 enrolled in the dose escalation portion of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Carotuximab (TRC105) Plus Capecitabine
Number analyzed (Participants) | 6
Participants
  Patients with DLT at 7.5 mg/kg | 0
  Patients without DLT at 7.5 mg/kg | 3
  Patients with DLT at 10 mg/kg | 0
  Patients without DLT at 10 mg/kg | 3

2. Secondary Outcome: TRC105 Steady State Pharmacokinetic Trough Concentration at the RP2D
Description: Mean trough concentration for patients dosed at 10 mg/kg at cycle 2 day 1
Time Frame: Cycle 2 day 1 (3 weeks)
Population: All patients who received full TRC105 doses of 10 mg/kg in cycle 1.
Measure: Mean (Full Range); unit: ng/mL
Groups:
- Single: All patients dosed at 10 mg/kg TRC105 who received TRC105 + capecitabine
  TRC105: IV (10 mg/kg weekly)
  Capecitabine: oral (1,000 mg/m2 BID)
Arm/Group | Single
Number analyzed (Participants) | 15
ng/mL | 66668.75 [200 to 129000]

3. Secondary Outcome: Number of Patients With Positive Immune Response to TRC105
Description: Serial blood samples will be tested for anti-drug antibody (ADA) immune response to TRC105. Patients who are positive at baseline (prior to receiving TRC105) are excluded from analysis.
Time Frame: 1.5 years
Population: All patients who received at least a portion of a dose of TRC105
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 19
Participants
  Post-Dose Positive Anti-Drug Antibody | 3
  Post-Dose Negative Anti-Drug Antibody | 16

4. Secondary Outcome: Number of Patients With Objective Response According to RECIST 1.1
Description: The best response according to RECIST 1.1 for each patient with measurable disease who received at least one dose of study drug will be listed by cohort and tumor type
Time Frame: 1.5 years
Population: Patients who had measurable disease at baseline and received at least one follow up scan were evaluable for the primary efficacy outcome of ORR by RECIST 1.1
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 16
Participants
  Partial Response | 1
  Stable Disease | 3
  Progressive Disease | 12

ADVERSE EVENTS:
Time Frame: Adverse events are collected for each patient from the time of informed consent through 28 days following the last dose of study drug. Patients were eligible for participation in the trial until they progressed. The longest duration of AE collection for a given patient was 1 year.
Arm/Group | Single
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 6/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single (N=19)
Fatigue (General disorders) | 1 (1) — Unrelated per investigator assessment to TRC105
Headache (Nervous system disorders) | 1 (1) — Suspected related to TRC105 per investigator assessment
Pyrexia (General disorders) | 1 (1) — Unrelated per investigator assessment to TRC105
Fracture (Injury, poisoning and procedural complications) | 1 (1) — Unrelated per investigator assessment to TRC105
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — Unrelated per investigator assessment to TRC105
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) — Unrelated per investigator assessment to TRC105
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single (N=19)
Headache (Nervous system disorders) | 7 (7) — Suspected related to TRC105 by the investigator
Fatigue (General disorders) | 7 (7) — Suspected related to TRC105 by the investigator
Gingival bleeding (Gastrointestinal disorders) | 7 (7) — Suspected related to TRC105 by the investigator
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) — Suspected related to TRC105 by the investigator
Vomiting (Gastrointestinal disorders) | 5 (5) — Suspected related to TRC105 by the investigator
Nausea (Gastrointestinal disorders) | 5 (5) — Suspected related to TRC105 by the investigator
Infusion-related reactions (Injury, poisoning and procedural complications) | 4 (4) — Suspected related to TRC105 by the investigator
Flushing (Vascular disorders) | 3 (3) — Suspected related to TRC105 by the investigator
Rash (Skin and subcutaneous tissue disorders) | 3 (3) — Suspected related to TRC105 by the investigator

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No